CLINICAL TRIAL: NCT00764192
Title: Angiologic Study of the Influence of Hemodialysis on Endothelial Function
Brief Title: Influence of Hemodialysis on Endothel-Depending Dilatation of Peripheral Arteries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Collaborators: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Christian Meyer, MD, RWTH Aachen University, Medical Clinic I, University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EK DD 2022 CM
Record Dates: First submitted 2008-09-26; First posted 2008-10-01 (Estimated); Last update posted 2009-01-13 (Estimated); Status verified 2009-01

CONDITIONS: Hemodialysis
Keywords: hemodialysis; Flow-mediated dilation; nictric oxide; endothelial function
MeSH Terms: interventions — Blood Specimen Collection; Lead

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 14 HD patients are studied before and after a single HD using a polysulphone dialyser.
  Interventions: Procedure: blood sample; Procedure: Flow-mediated dilation (FMD) before and after a single HD

INTERVENTIONS:
Procedure: blood sample — blood sample before and after a single HD
  Other Names: biochemistry
Procedure: Flow-mediated dilation (FMD) before and after a single HD — measuring of the flow-mediated dilation using high-resolution ultrasound
  Other Names: endothelial function

SUMMARY:
An impairment of nitric oxide (NO) bioavailability is associated with endothelial dysfunction and may contribute to the excessive incidence of cardiovascular complication in chronic haemodialysis (HD) patients. It is not known whether cell-free hemoglobin limits nitric oxide bioavailability during HD.

DETAILED DESCRIPTION:
Cardiovascular complications are the major cause of death in end-stage renal disease (ESRD) patients undergoing chronic haemodialysis (HD).1 During haemodialysis (HD) the endothelium is the first organ to sense and to be impaired by mechanical and immunological stimuli.2 Adequate endothelial function and integrity reduce thromboembolic events, while endothelial dysfunction is an early key step in the development of atherosclerosis3-5, is involved in plaque progression6 and has been attributed to impaired nitric oxide (NO) bioactivity and enhanced formation of oxygen-derived free radicals.7 Given that endothelial dysfunction is at least in part reversible, the assessment of altered NO availability is of important diagnostic and prognostic significance and may deepen the understanding of cardiovascular disease in HD.8 Nitric oxide bioavailability has been shown to be limited by cell-free hemoglobin.9 The rates of NO consumption by cell-free and intraerythrocytic hemoglobin suggest that only when hemoglobin is physically compartmentalized within erythrocytes will NO produced by endothelial cells reach concentrations within smooth muscle necessary to activate guanylyl cyclase and cause vasodilation.10;11 However, the rate of NO scavenging is reduced 1,000-fold by sequestering hemoglobin within the red cell membrane.12;13 This mechanism is believed to be important in various conditions of health and disease.14-16 In ESRD intravascular hemolysis during HD has been described.17-19

ELIGIBILITY:
Inclusion Criteria:

* patients older 21 years dependent on HD for more than 6 months

Exclusion Criteria:

* known HD associated hypotension intake of nitrate

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-10; Primary Completion 2007-02 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
influence of hemodialysis on endothelial function as determined by plasma nitrite concentration | before and after hemodialysis

SECONDARY OUTCOMES:
influence on hemodialysis on endothelial function as determined by measurement of flow-mediated dilation (FMD) of teh brachial artery using high resolution ultrasound | before and after hemodialysis

CONTACTS AND LOCATIONS:
Overall Officials: Christian Meyer, MD, Principal Investigator — RWTH Aachen University, Medical Clinic I
Locations (1):
- University Hospital, Aachen, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Meyer C, Heiss C, Drexhage C, Kehmeier ES, Balzer J, Muhlfeld A, Merx MW, Lauer T, Kuhl H, Floege J, Kelm M, Rassaf T. Hemodialysis-induced release of hemoglobin limits nitric oxide bioavailability and impairs vascular function. J Am Coll Cardiol. 2010 Feb 2;55(5):454-9. doi: 10.1016/j.jacc.2009.07.068. PMID 20117459